CLINICAL TRIAL: NCT03282968
Title: Balance Training With the Rehabilitative Wayout In Responsive Home Environments (REWIRE) System in Patients After Stroke
Brief Title: Balance Training After Stroke With REWIRE
Acronym: REWIRESI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Collaborators: Jozef Stefan Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: URIS201704
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: exergaming; physiotherapy; balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Regular neurophysiotherapy plus REWIRE exercises
  Interventions: Device: REWIRE
- Control (Active Comparator): Regular neurophysiotherapy plus standing balance exercises
  Interventions: Other: Balance exercises

INTERVENTIONS:
Device: REWIRE — First, the patient will play the Fruit Catcher (weight transfer) game on the 3rd level for 3 minutes, followed by 3 minutes of rest. Next, the patient will play the Horse Runner (squats) on the 3rd level for 3 minutes, followed by 3 minutes of rest. In the end, the patient will play the Animal Hurdler (standing on one leg) on the 3rd level for 3 minutes. During the games, the patient will be standing on the Wii Balance Board, holding to a firm support if necessary. During the rest periods, the patients will be sitting. A physiotherapist will be present throughout the exercise for safety and help if requested.
  Arms: Experimental
Other: Balance exercises — The patient will first practice balance transfer for 3 minutes (standing by a ladder, holding position on each leg for 3 seconds), followed by 3 minutes of rest. Next, the patient will be performing squats for 3 minutes, followed by 3 minutes of rest. In the end, the patient will practice alternatively lifting lower limbs (like stepping on a footstool) for 3 minutes. During the rest periods, the patients will be sitting. A physiotherapist will be present throughout the exercise for safety and help if requested.
  Arms: Control

SUMMARY:
The study will include 20 patients after stroke, randomly assigned to the experimental and control group (10 each). In both groups, the program with last for five days; walking and balance will be assessed before and after the program. Both groups will receive regular neurophysiotherapy; in addition, the experimental group will exercise each day by playing REWIRE games, while the control group will perform standing balance exercises.

DETAILED DESCRIPTION:
Detailed inclusion and exclusion criteria are specified in the appropriate section. Both groups will perform the additional exercises for 15 minutes daily. In addition to the outcome measurement, informal feedback will be obtained from the patients and the therapists on the feasibility of the REWIRE system.

ELIGIBILITY:
Inclusion Criteria:

* first stroke
* first admission to inpatient rehabilitation

Exclusion Criteria:

* less than 25 points scored on the Mini-Mental State Examination
* inability to walk independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in walking speed | Assessment one day before and one day after the program
  Assessed using 10 Meter Walking Test
Change in dynamic balance | Assessment one day before and one day after the program
  Assessed using Four Step Square Test

SECONDARY OUTCOMES:
Change in mobility | Assessment one day before and one day after the program
  Assessed using Timed Up and Go test
Change in static standing balance | Assessment one day before and one day after the program
  Assessed using Romberg test

CONTACTS AND LOCATIONS:
Overall Officials: Imre Cikajlo, PhD, Principal Investigator — University Rehabilitation Institute, Rehabilitation of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cikajlo I, Rudolf M, Mainetti R, Borghese NA. Multi-Exergames to Set Targets and Supplement the Intensified Conventional Balance Training in Patients With Stroke: A Randomized Pilot Trial. Front Psychol. 2020 Apr 2;11:572. doi: 10.3389/fpsyg.2020.00572. eCollection 2020. PMID 32300321